CLINICAL TRIAL: NCT02597946
Title: A Phase II Study of Afatinib in Patients With Advanced NSCLC Harboring HER2 Mutations, Previously Treated With Chemotherapy
Brief Title: Afatinib in NSCLC With HER2 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.222
Record Dates: First submitted 2015-11-02; First posted 2015-11-05 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Paclitaxel

ARMS (1):
- all patients (Experimental): Part A: all enrolled patients will receive afatinib monotherapy. Part B: all eligible patients will receive afatinib combined with weekly paclitaxel.
  Interventions: Drug: afatinib; Drug: paclitaxel

INTERVENTIONS:
Drug: afatinib
Drug: paclitaxel

SUMMARY:
to investigate effectiveness and safety of afatinib in the advanced NSCLC patients with HER2 mutations, previously treated with 1 or 2 chemotherapy regimens

ELIGIBILITY:
Inclusion criteria:

* Patients with Histologically or cytologically confirmed diagnosis of stage IIIb/IV NSCLC (AJCC 7.0), who had failed one or two systemic chemotherapy regimens, one of which must be platinum-based .
* Tumor tissue with HER2 mutations as confirmed by AmoyDx® HER2 Mutation Detection Kit
* Patients with at least one measurable tumor lesion that can accurately be measured by CT scan or MRI according to RECIST 1.1
* Age>=18 years
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
* Adequate organ function
* Recovered from any previous therapy related toxicity to <=Grade 1 at study entry (except for stable sensory neuropathy <=Grade 2 and alopecia)
* Written informed consents that is consistent with International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP) and local GCP guidelines Inclusion criterion for Part B
* Adequate organ function, as inclusion criteria No.6
* ECOG performance score 0~2
* More than 12 weeks clinical benefit (PR, Complete Response (CR), SD) in part A Further inclusion criteria apply

Exclusion criteria:

* Prior treatment with Epidermal Growth Factor Receptor (EGFR) or HER2 targeting small molecules or antibodies.
* Any chemo-, or immune anticancer therapy within 4 weeks prior to start of study treatment, Hormonal treatment within 2 weeks prior to start of study treatment, Radiotherapy within 4 weeks prior to start of treatment, except as follows:

  i.) Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to enter, and ii.) Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
* Known hypersensitivity to afatinib or the excipients of any of the trial drugs
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of >= 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug.
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Requiring treatment with any of the prohibited concomitant medications
* Known pre-existing interstitial lung disease.
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug.
* Active hepatitis B infection and/or active hepatitis C infection and/or known HIV carrier.
* Leptomeningeal carcinomatosis.
* Symptomatic brain metastases; To be eligible patients must be asymptomatic from brain metastases at least 4 weeks without requirement for steroids or anti-epileptic therapy.
* Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control for the duration of study participation and for at least 2 weeks after treatment has ended.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial Exclusion criterion for Part B Any known contraindication for paclitaxel treatment. Not able to tolerate lowest dose of afatinib. Peripheral polyneuropathy >Grade 2 Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (9):
- China (8):
  - Hunan Province Tumor Hospital, Changsha
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - First Hospital Affiliated with Nanjing Medical University, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Henan Cancer Hospital, Zhengzhou
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open label, single arm study, divided into 2 parts; Part A: All enrolled patients will receive afatinib monotherapy.Part B: Patients with more than 12 weeks clinical benefit in part A will receive afatinib once daily combined with paclitaxel once weekly.
Pre-assignment Details: No patients met the criteria to enter part B. Thus part B was not performed in this trial.
Groups:
- Afatinib 40 mg (Part A): Patients were orally administered 40 milligram (mg) Afatinib film-coated tablets daily starting dose, once daily continuous (possible escalation to 50 mg, and reduction to 30 mg in the first step, and to 20 mg in the second step) until disease progression or intolerable toxicity or withdrawal of consent for any reason.
Period: Overall Study
Arm/Group | Afatinib 40 mg (Part A)
Started | 18
Completed | 0
Not Completed | 18
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 16
Not completed — Other than above | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Treated set included all patients who were documented to have taken at least 1 dose of afatinib
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Objective Response (OR) in Part A According to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1
Description: Percentage of patients with objective response (OR) in part A according to RECIST 1.1. Objective Response defined as patients with tumour size reduction of a predefined amount using RECIST 1.1 in part A. Objective response included both confirmed Partial Response (PR) plus Complete Response (CR) as measured by Computed Tomography (CT) scan or Magnetic Resonance Imaging (MRI) according to RECIST 1.1.
  Partial Response (PR): At least a 30% decrease in the sum of longest diameter (LD) of target lesions asking as reference the baseline sum LD. Complete Response (CR): Disappearance of all target lesions.
Time Frame: CT Scan at Weeks 8 & 12 (for week 12 tumor assessment, time window is +1week), then every 8 weeks thereafter, after week 52, assessments will be performed every 12 weeks until progression or start of further treatment , ie., up to approximately 12 Months
Population: Treated Set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 18
Percentage of participants | 0.0

2. Secondary Outcome: Percentage of Patients With Disease Control (DC) in Part A
Description: Percentage of patients with disease control (DC) in part A. Disease control defined as patients who have achieved confirmed complete response, partial response and stable disease as measured by CT scan or MRI according to RECIST 1.1 in part A.
  Tumour Response is based on clinical, radiological or other assessment. Clopper-Pearson method used for confidence limits.
  Partial Response (PR): At least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. Complete Response (CR): Disappearance of all target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR, taking as reference the baseline sum LD, nor sufficient increase to qualify for Progression (PD) taking as reference the smallest sum LD since the treatment started.
Time Frame: CT Scan at Weeks 8 & 12(for week 12 tumor assessment, time window is +1week), then every 8 weeks thereafter, after week 52, assessments will be performed every 12 weeks until progression or start of further treatment, ie up to approximately 12 Months
Population: Treated set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 18
Percentage of participants | 61.1 [35.7 to 82.7]

3. Secondary Outcome: Progression Free Survival (PFS) in Part A
Description: Progression Free Survival (PFS) defined as the time from the date of starting treatment of afatinib to the date of disease progression per RECIST 1.1, or to the date of death no matter which happens first in part A.
  Median and 95% confidence interval (CI) are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From the date of starting treatment of afatinib to the date of disease progression or to the date of death, ie up to approximately 12 Months
Population: Treated set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 18
Months | 2.76 [1.87 to 4.60]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) defined as the time from start of treatment of afatinib until death from any cause.
  Median and 95% CI are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From start of treatment of afatinib until death from any cause, ie up to approximately 12 Months
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 18
Months | 10.02 [8.47 to 10.08]

5. Secondary Outcome: Time to Progression (TTP) in Part A
Description: Time to progression (TTP) defined as the time from the date of starting treatment of afatinib to the date of disease progression per RECIST 1.1 in part A.
  Median and 95% CI are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From the date of starting treatment of afatinib to the date of disease progression , ie up to approximately 12 Months
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 18
Months | 2.76 [1.87 to 4.60]

6. Secondary Outcome: Duration of Response (DOR) in Part A
Description: Duration of response (DoR) defined as the time from the first documented response PR or CR to the date of tumor progression evaluated according to RECIST 1.1 or death in part A.
  Partial Response (PR): At least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. Complete Response (CR): Disappearance of all target lesions.
  No patient had objective response and DoR was not analysed.
Time Frame: as for outcome 2
Population: No patient had objective response and DoR was not analysed.
Arm/Group | Afatinib 40 mg (Part A)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after the last dose, ie up to 272 days.
Arm/Group | Afatinib 40 mg (Part A)
All-Cause Mortality (participants affected / at risk) | 8/18
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (Part A) (N=18)
Gastroenteritis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Thrombosis (Vascular disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Malaise (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (Part A) (N=18)
Upper respiratory tract infection (Infections and infestations) | 3
Paronychia (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Myringitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Influenza like illness (General disorders) | 1
Pyrexia (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 12

LIMITATIONS AND CAVEATS:
No patients met the criteria to enter Part B. Thus planned Part B was not performed in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02597946/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02597946/SAP_000.pdf